CLINICAL TRIAL: NCT07403708
Title: Retromandibular Transparotid Approach Versus Transmasseteric Anteroparotid Approach for Fixation of Subcondylar Fracture: Randomized Controlled Clinical Study
Brief Title: Retromandibular Transparotid Approach Versus Transmasseteric Anteroparotid Approach for Fixation of Subcondylar Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, mona oraby, Dr., Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0841-01/2024
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Condylar Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transmasseteric anteroparotid approach (Experimental)
  Interventions: Procedure: transmasseteric anteroparotid approach
- transparotid approach (Active Comparator)
  Interventions: Procedure: transparotid approach

INTERVENTIONS:
Procedure: transmasseteric anteroparotid approach — safer approach for condylar fracture
  Arms: transmasseteric anteroparotid approach
Procedure: transparotid approach — facial nerve and parotid dissection to reach condyle
  Arms: transparotid approach

SUMMARY:
Background: Condylar fracture is one of mandibular fracture which accounts for 20-35%. It is the most controversial fractures regarding diagnosis and management. For several years, surgeons preferred closed reduction over open reduction to avoid surgical complications.

Closed reduction may have late complications, the preference started to change towards open treatment. A Transmasseteric Anteroparotid (TMAP) approach for open treatment of condylar fractures overcomes the problems of facial nerve injury of other approaches. Aim: Comparing the Transmasseteric Antroparotid approach(TMAP) to the Transparotid (TP) approach in management of subcondylar fractures regarding the facial nerve affection, parotid fistula, reduction angulation, pain, duration of the surgery, occlusion and patient satisfaction with the scar. Materials and Methods: Twenty patients with subcondylar fracture will be divided randomly into two equal groups. Group1(study group): Transmasseteric Antroparotid approach. Group2 (control group): Retromandibular Transparotid approach. Patients will be followed up for 3 months to assess facial nerve injury, pain, occlusion and patient's scar satisfaction . Results: data will be collected, tabulated and statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from displaced extracapsular mandibular subcondylar fracture indicated for open reduction including:

Difficulty of obtaining adequate occlusion by closed method. Radiological signs of the following:

1. Deviation of the he fragments from the axis of the ascending ramus in medial or lateral direction more than 10°. (28)
2. Shortening of the ascending ramus ≥ 2 mm measured from the roof of glenoid fossa to the inferior border of the ascending ramus of the mandible.
3. Dislocation of the condyle from the glenoid fossa.

Exclusion Criteria:

* Patients who were not able to follow the information given or to make a decision themselves due to mental or other problems. 2. Patient with undisplaced condylar fractures that doesn't cause malocclusion or loss of facial heightening and can be treated conservatively.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
facial nerve injury | immediate postoperative

SECONDARY OUTCOMES:
approach time | interaoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No